CLINICAL TRIAL: NCT05139212
Title: An Optimum Time for Intravenous Cannulation After General Anesthesia Induction With Sevoflurane and Nitrous Oxide in Children Undergoing Elective Surgery With Dexmedetomidine Premedication
Brief Title: Determination of Optimum Time for Intravenous Cannulation in Children With Dexmedetomidine Premedication
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 08-2021/02
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-11

CONDITIONS: Cannulation; Sevoflurane Induction; Dexmedetomidine
Keywords: Induction of anesthesia; Sevoflurane; Nitrous oxide; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Procedure: Optimum time for intravenous cannulation in children premedicated with dexmedetomidine — The optimum time for intravenous cannulation after the induction of anesthesia with sevoflurane, oxygen, and nitrous oxide in children with intranasal dexmedetomidine premedication will be searched in children undergoing elective surgery.

SUMMARY:
Inhalational induction with sevoflurane, nitrous oxide, and oxygen is accepted as a safe technique to avoid any movement during intravenous cannulation in children. In addition, intranasal dexmedetomidine could be used for premedication to reduce preoperative anxiety in preschool children. Early attempts to place, an intravenous line may result in movement and respiratory complications like coughing or laryngospasm. On the other hand delay in cannulation may prevent effective management of bradycardia and hypotension. There are a number of studies examining the optimum time for cannulation after sevoflurane induction. However, it is not known whether the addition of dexmedetomidine premedication affects the time for intravenous cannulation following induction with sevoflurane and nitrous oxide.

DETAILED DESCRIPTION:
All the children will be premedicated with intranasal 2mcg/kg dexmedetomidine 40 minutes before the surgery. Ramsay sedation scale and Turkish version of modified Yale Preoperative Anxiety Scale (mYPAS) will be measured at the time of arrival in the daycare unit and during anesthesia preparation in the operating room.

The same anesthesia machine will be used in all children with the same circuit volume. The circuit will be emptied and then filled with sevoflurane (8%) and nitrous-oxygen (50:50) for 30 seconds at a high fresh gas flow (6 liter/minute). The timer will be started when the face mask is placed on the child's face for inhalational induction.

The exhaled gas concentrations will be measured continuously. After the loss of eyelash reflex, the fresh gas flow will be reduced to 3 liter/minute, the sevoflurane will be reduced to 5% and the timer will be restarted. Spontaneous respiration will be allowed until intravenous cannulation and ventilation will be gently assisted as required.

For the first child, the gas flow settings will be maintained for 4 minutes from the loss of eyelash reflex before intravenous cannulation is attempted. All intravenous cannulation will be performed on the dorsum of the hand by an experienced anaesthesiologist, using a 24-gauge stainless steel guide cannula.

At the time of intravenous cannulation attempt, an independent observer, who will be blinded about the predetermined cannulation time, will rate the movement according to a scale (0= no movement, 1= slight extremity tension, 2= extremity withdrawal, 3= generalized movement).

The intravenous cannulation will be considered unsuccessful if there is any movement, cough, or laryngospasm, and the procedure will be considered successful in the absence of any reaction.

The time for the subsequent patient's intravenous cannulation will be adjusted accordingly using Dixon's up-down sequential method (starting at 4 min with 15 s as the step size). The time for cannulation will be increased by 15 s if the time will be inadequate in the previous patient, and conversely, the time for cannulation will be decreased by 15 s if the time will be adequate in the previous patient.

The aim of this study will be to determine the optimum time for intravenous cannulation after the induction of anesthesia with sevoflurane, oxygen, and nitrous oxide in children with intranasal dexmedetomidine premedication.

ELIGIBILITY:
Inclusion Criteria:

* Children with ASA physical status I and scheduled for an elective procedure under general anesthesia without prior intravenous cannulation will be selected

Exclusion Criteria:

* Children posted for any emergency procedure
* ASA class II and above,
* Children with abnormal airway anatomy.
* Children with active respiratory infection in the last 3 weeks.
* Children who are being treated with sedative or anticonvulsive agents.
* Children with heart, lung, neurologic, or central nervous system disorders.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 2-6 years, American Society of Anesthesiologists physical status 1 scheduled for elective procedures undergoing inhalational induction after dexmedetomidine premedication without intravenous access will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Determination of optimum time for intravenous cannulation after induction with sevoflurane and nitrous oxide in children premedicated with dexmedetomidine | The outcome will be assessed at the time of intravenous cannulation attempt.
  At the time of intravenous canulation attempt, an independent observer who will be blinded about predetermined canülation time, rated the movement according to a scale (0= no movement 1= slight extremity tensing, 2= extremity withdrawal, 3=generalized movement.
  Intravenous cannulation without any laryngospasm or movement will be considered successful.

SECONDARY OUTCOMES:
To assess level of preoperative sedation | Assesment of children will be started from acceptance of patient to preoperative holding area to the time of anesthesia preparation.
  The level of sedation will be assessed with Ramsay Sedation Scale. This scale includes the following categories: 1, anxious, restless, or agitated; 2, cooperative; 3, responds to commands only; and 4-6, different levels of unconsciousness, where 6 indicates no response to a light glabellar tap or loud auditory stimulus. Higher scores denote higher levels of sedation. Assessment will be started from acceptance of the patient to the preoperative holding area (baseline) to the time when anesthesia preparation will occur. The children will be evaluated 3 times, at baseline, post-premedication 40th minute, and during anesthesia preparation in the operating room.
To assess level of preoperative anxiety | Assesment of children will be started from acceptance of patient to preoperative holding area to the time of anesthesia preparation.
  Anxiety will be measured at the time of arrival in the preoperative holding area (baseline) and during anesthesia preparation in the operating room. The level of anxiety will be assessed using the validated Turkish version of the modified Yale Preoperative Anxiety Scale (mYPAS), containing 27 items in five categories (activity, emotional, expressivity, state of arousal, vocalization, and use of parents), representing five domains ofanxiety.The mYPAS scale ranges from 0 to 100 points, with higher scores signifying higher levels of anxiety. Assessment will be started from acceptance of the patient to the preoperative holding area (baseline) to the time when anesthesia preparation will occur. The children will be evaluated 3 times, at baseline, post-premedication 40th minute, and during anesthesia preparation in the operating room.

CONTACTS AND LOCATIONS:
Overall Officials: Rafet Yarimoglu, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Taining and Research Hospital, Karaman, Turkey (Türkiye)